CLINICAL TRIAL: NCT03724344
Title: Correlation Analysis Between Mental Behavioral Symptoms in Dementia Patients and Mood Disorders of Caregivers
Brief Title: Correlation Study Between Mental Behavioral Symptoms in Dementia Patients and Mood Disorders of Caregivers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: HKM201721
Record Dates: First submitted 2018-10-27; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2017-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dimensions with Behavioral and psychological symptoms
  Interventions: Other: Cross section resaerch

INTERVENTIONS:
Other: Cross section resaerch — Assessment of cognitive (MoCA), mental behavioral symptoms (NPI） the Self-rating Depression Scale (SDS) and the Self-rating Anxiety Scale (SAS).

SUMMARY:
Traditionally, the more severity of dementia patients, the heavier the burden of the comparators, and in the clinical observation,the dementia patients with rich mental behavior symptoms are more burdened. Therefore, exploring the impact of psychological burden and different subtypes of different dimensions with Behavioral and psychological symptoms (BPSD) will more comprehensive understanding of the factors affecting the burden of caregivers.

The starting point of this project is to analyze the relationship between the types of mental behavior symptoms of dementia patients and the emotional disorders of caregivers. The topic will analyze the correlation of psychological burden of caregivers and different symptom dimensions from the perspective of refinement, helping more effective identifying high-burden mental behavior symptoms in clinically , judging the risk of emotional problems in caregivers, and adopting better humanities or medical care, so that dementia patients can better adapt to care and improve the mental health of caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. Age is greater than 18 years old, gender is not limited
2. Comply with ICD-10 diagnostic criteria, diagnosed with dementia, including Alzheimer's disease, vascular dementia, frontotemporal dementia, dementia with Lewy body, dementia caused by Parkinson's disease

Exclusion Criteria:

1. senile schizophrenia;
2. senile depression;
3. cognitive impairment caused by endocrine system diseases (such as decreased thyroid and adrenal function);
4. Cognitive impairment or dementia caused by serious diseases such as cardiovascular, lung, liver, kidney, and hematopoietic system;
5. Cognitive impairment or dementia caused by alcohol, drug use, psychotropic drugs; 6）Other physical or chemical factors that cause cognitive impairment or dementia-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Outpatients and community dementia patients and their primary caregivers
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric inventory questionnaire | baseline
  Behavioral and psychological symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Zhenghui Yi, MD, Study Chair — Shanghai Mental Health Center
Locations (1):
- Huangpu District Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No